CLINICAL TRIAL: NCT00572949
Title: Magnetocardiography (MCG) in the Diagnosis of Chest Pain Syndrome
Status: Withdrawn | Type: Observational
Why Stopped: sponsor funding
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: CardioMag Imaging (Industry)
Responsible Party: Kirsten Tolstrup,MD, Cedars-Sinai Medical Center
Other Study IDs: 4039
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2009-11-17 (Estimated); Status verified 2009-11

CONDITIONS: Chest Pain
Keywords: heart disease; chest pain; coronary artery disease; atherosclerosis
MeSH Terms: conditions — Chest Pain; Heart Diseases; Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with chest pain syndrome

SUMMARY:
The purpose of this research study is to evaluate a better way of diagnosing heart artery disease, heart attack and damage to the heart muscle early on. Currently, it often takes several hours after admission before lab tests will show that there has been any damage to the heart muscle. Although the standard electrocardiogram is quick and non-painful it may miss many cases of significant coronary heart disease. The investigators are proposing that a new entirely non-contact tool, the Magnetocardiograph (MCG), with high accuracy is able to predict the presence of significant coronary heart disease early on before other studies become positive. The investigators hope by this that the investigators can develop an algorithm for better triage and management of patients with chest pain.

This research study is designed to test the effectiveness of the investigational use of the Magnetocardiograph (MCG) that has been approved by the U.S Food and Drug Administration (FDA). While the MCG used in the study is FDA-approved as a tool for the non-contact measurement and display of the magnetic fields of the heart generated by the electrical currents, it is not yet approved for the specific diagnosis of heart artery disease (ischemia).

DETAILED DESCRIPTION:
Cardiomagnetism refers to the detection, analysis and interpretation of the magnetic fields generated by the electrical activity of the heart. The peak value of the magnetic fields of the heart is more than a million times smaller than the Earth's magnetic field. A major breakthrough in the capability of measuring such small fields came with the invention of the SQUID (superconducting quantum interference device) in the late sixties. The first magnetocardiograms (MCGs) measured with the SQUID were recorded by Cohen et al. in 1970 (1). These earlier measurements were performed in very expensive magnetically shielded rooms, initially utilizing only one or two SQUID probes. In the eighties this technology was tested in several laboratories creating a magnetic field map by moving one SQUID sequentially above the chest to create an image of the whole hearts magnetic field. These maps were then attempted correlated with various pathologies (2,3).

Since then the technology has been greatly improved and several multichannel machines are in use across the world for research purpose for arrhythmia localization and ischemia detection. However, at present time, only one company (CardioMag Imaging) has developed a machine that operates outside a shielded room.

The CardiomagImaging (CMI) Magnetocardiograph (MCG) is capable of noninvasive recording of magnetic fields arising from the electrical activity of the heart with very high spatial and temporal resolution. The temporal trace of the MCG is analogous to an ECG, and, similarly, can be recorded in multiple leads. This MCG device has been specifically developed for the general purpose (outside shielded room) of non-contact, non-invasive diagnostics of ischemia.

The CMI MCG device has been approved as safe for patients. It is FDA approved for the noninvasive detection and display of the heart's magnetic field created by the electrical currents, and is awaiting FDA approval for the detection of ischemia in chest pain patients. A similar SQUID technology utilized in magnetically shielded rooms has already been FDA approved for localization of epileptic focus. When utilized in this matter it is referred to as MEG (magnetoencephalogram).

Several abstracts have been presented primarily at meetings on Biomagnetism, that confirm the safety and indicate the efficacy of the MCG for the detection of ischemia. In particular, it has been suggested that the resting MCG is capable of detecting ischemia in patients with chest pain, when the 12-leads ECG is normal (4,5,6). However, this has not been tested in larger prospective blinded studies.

Cedars-Sinai Medical Center Non-invasive Cardiac Laboratory will be the first center in the US evaluating the CardioMag Imaging MCG in a clinical environment for the detection of ischemia in an acute coronary syndrome patient population. Patients will be enrolled in a similar protocol at Johns Hopkins Medical Center, Baltimore, Mayo clinic, Rochester, and at Klinikum Hoyerswerda, Germany. The early detection of ischemia (before Troponins become positive) with high negative and positive predictive values may prove cost effective and decrease risk by improving prompt treatment and triage to higher or lower grade monitoring at time of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chest pain syndrome

Exclusion Criteria:

* ST elevation MI
* Hemodynamically unstable patients
* Tachycardia with heart rate >150 just prior to testing or at time of testing
* A-V Dissociation on 12-lead ECG
* Patients with pacemakers or internal defibrillators
* Minors < 18 years of age
* Patients unable to lie flat for the examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chest pain syndrome
Sampling Method: Probability Sample
Enrollment: 398 (Estimated)
Dates: Start 2004-10; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Tolstrup, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] 1) Cohen D, Edelsack EA, Zimmerman JE. Magnetocardiograms taken inside a shielded room with a superconducting point-contact magnetometer. Appl. Phys. Lett. 1970, 16, 278-280.
- [Background] Nakaya Y, Sumi M, Saito K, Fujino K, Murakami M, Mori H. Analysis of current source of the heart using isomagnetic and vector arrow maps. Jpn Heart J. 1984 Sep;25(5):701-11. doi: 10.1536/ihj.25.701. PMID 6239932
- [Background] 3) Stroink G, MacAuley C, Montague TJ, Horacek BM. Normal and abnormal components in magnetocardiographic maps of a subject with myocardial infarction. Med. Biol. Eng. Comp. 1985, 23, 61-62.
- [Background] 4) Brazdeikis A, Taylor AA, Mahmarian JJ, Xue Y, Chu CW. Comparison of magnetocardiograms acquired in unshielded clinical environment at rest, during and after exercise and in conjunction with myocardial perfusion imaging. Biomag 2002, 530-532.
- [Background] 5) Chaikovsky I, Primin M, Nedayvoda I, Vassylyev V, Sosnitsky V, Steinberg F. Computerized classification of patients with coronary artery disease but normal or unspecifically changed ECG and healthy volunteers. Biomag 2002, 534-536.
- [Background] Morguet AJ, Behrens S, Kosch O, Lange C, Zabel M, Selbig D, Munz DL, Schultheiss HP, Koch H. Myocardial viability evaluation using magnetocardiography in patients with coronary artery disease. Coron Artery Dis. 2004 May;15(3):155-62. doi: 10.1097/00019501-200405000-00004. PMID 15096996